CLINICAL TRIAL: NCT03523936
Title: Gut Microbiota and Antibiotics - Prevention of Side Effects by New Prebiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: VTT Technical Research Centre of Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T63/2018
Record Dates: First submitted 2018-05-02; First posted 2018-05-14 (Actual); Last update posted 2018-05-14 (Actual); Status verified 2018-05

CONDITIONS: Changes in the Gut Microbiota During an Antibiotic Treatment
Keywords: antibiotics, prebiotics, dysbiosis
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prebiotic (Active Comparator)
  Interventions: Dietary Supplement: Prebiotic product
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic product — Prebiotic product used during the course of antibiotic treatment
  Arms: Prebiotic
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Antibiotics disturb the balance of gut microbiota causing dysbiosis. The purpose of this double-blind placebo controlled intervention study is to investigate whether a new prebiotic product could prevent the side effects of antibiotics.

DETAILED DESCRIPTION:
Thirty children (2-6 years of age), who require antibiotic treatment assessed by a doctor, will be enrolled in the study. The children will be randomized to receive either the prebiotic product or placebo during the course of antibiotic treatment.

The children will give a faecal sample in the beginning and at the end of the study. The samples will be used for the analysis of microbiota and differences in the microbiota between the groups.

ELIGIBILITY:
Inclusion Criteria:

* An infection requiring antibiotic treatment assessed by a doctor

Exclusion Criteria:

* Coaeliac disease or allergy to cereals, use of other prebiotic/probiotic product during the study

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of gut microbiota during antibiotic treatment | One week
  Gut microbiota and antibiotics - Prevention of side effects by new prebiotics